CLINICAL TRIAL: NCT02023788
Title: Long-term Safety and Efficacy Follow-up Study of PNEUMOSTEM® in Patients Who Completed PNEUMOSTEM® Phase-I Study
Status: Completed | Type: Observational
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MP-CR-006-F/U-5y
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2017-04

CONDITIONS: Bronchopulmonary Dysplasia; Respiratory Tract Infections; Premature Birth of Newborn
Keywords: human umbilical cord blood-derived mesenchymal stem cells; bronchopulmonary dysplasia; respiratory tract infection; Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Tract Infections; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pneumostem®: Low Dose Group (3 subjects): 1.0 x 10^7 cells/kg, High Dose Group (6 subjects): 2.0 x 10^7 cells/kg
  Intervention: Biological: Pneumostem®
  Interventions: Biological: PNEUMOSTEM

INTERVENTIONS:
Biological: PNEUMOSTEM — A single intratracheal administration
  Low Dose Group (3 patients): 1.0 x 10^7 cells/kg High Dose Group (6 patients): 2.0 x 10^7 cells/kg
  * The subjects were administered with Pneumostem in the earlier part of the Phase I study. No drug/biologics will be administered to any subject during this part of the study.
  Other Names: human umbilical cord blood-derived mesenchymal stem cells

SUMMARY:
This is a 5-year long-term follow-up study of open label, single-center, phase I clinical trial to evaluate the safety and efficacy of PNEUMOSTEM® in premature infants with bronchopulmonary dysplasia.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is the most common cause of death for prematurely born babies with low birth weights. In addition, many children who recover from this disease suffer from various complications such as prolonged hospitalization, pulmonary hypertension, and failure to thrive.

It has been reported that bone marrow-derived mesenchymal stem cells (BM-MSC) can differentiate into pulmonary epithelial and pulmonary endothelial cells. Some animal studies showed that BM-MSCs differentiate into bronchial cells and type 2 pneumocytes in rats with pneumonia and improve the fibrosis that occur after administration of bleomycin. Based on the findings, it is considered that mesenchymal stem cell therapy can help regenerate the damaged lung as well as BPD that cause lung inflammation, fibrosis, deficiency of type 2 pneumocytes, and so on.

PNEUMOSTEM® consists of human umbilical cord blood-derived mesenchymal stem cells and is intended to treat BPD in premature infants. The purpose of the study is to evaluate 3-5 year long term safety and efficacy in patients who completed the earlier part of the phase I clinical trial of PNEUMOSTEM®.

ELIGIBILITY:
Inclusion Criteria:

* All infants who were enrolled in the 2-year follow-up study (NCT01632475) of phase 1 clinical trial for the safety and efficacy evaluations of PNEUMOSTEM® treatment in premature infants with bronchopulmonary dysplasia
* Infants with a written consent form signed by a parent or legal guardian

Exclusion Criteria:

-Infants whose parent or legal guardian does not consent to participate in this follow-up study

Ages: 45 Months to 63 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who were enrolled in the 2-year follow-up study (NCT01632475) of phase 1 clinical trial for the safety and efficacy evaluations of PNEUMOSTEM® treatment in premature infants with bronchopulmonary dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse drug reactions | 60 months (corrected age)
  adverse drug reactions, clinically significant laboratory findings, vital signs, physical exam

SECONDARY OUTCOMES:
Respiratory outcomes | 60 months (corrected age)
  * hospital readmission rates and length of stay
  * whether medical interventions such as oxygen, steroid, or bronchodilator therapy was done and duration of the therapy
  * Frequency of Emergency Room visit (total number of visits/ number of visits due to respiratory illnesses)
Survival | 60 months (corrected age)
Z-score | 60 months (corrected age)
  * weight
  * height
  * head circumference
  * percentile
Potential neurological development test outcomes | 60 months (corrected age)
  * K-ASQ (Korean Ages and Stages Questionnaires),
  * Bayley test (BSID III)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Soon Park, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- See also: Phase-I: 2 Year Follow-Up Safety and Efficacy Study of Pneumostem® in Premature Infants With Bronchopulmonary Dysplasia — http://www.clinicaltrials.gov/ct2/show/record/NCT01632475?term=pneumostem&rank=1
- See also: Phase-I:Safety and Efficacy Evaluation of PNEUMOSTEM® Treatment in Premature Infants With Bronchopulmonary Dysplasia — http://www.clinicaltrials.gov/ct2/show/NCT01297205?term=pneumostem&rank=4
- See also: Phase-II: Efficacy and Safety Evaluation of Pneumostem® Versus a Control Group for Treatment of BPD in Premature Infants — http://www.clinicaltrials.gov/ct2/show/NCT01828957?term=pneumostem&rank=2